CLINICAL TRIAL: NCT06425458
Title: Transitioning Youth Out of Homelessness 2.5: A Co-Designed Strengths-Based Leadership Program for Young People Transitioning Out of Homelessness
Brief Title: Transitioning Youth Out of Homelessness 2.5 (TYOH 2.5)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Covenant House Toronto (Other); StepStones for Youth (Unknown); Resource Association for Teens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-072
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Homelessness; Youth
Keywords: Identity Capital; Youth; Coach; Self-Efficacy; Self-Esteem; Control; Purpose; Socioeconomic Inclusion; Homelessness; Transition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Co-Designed Strengths-Based Leadership Program (Experimental): Young people transitioning out of homelessness will attend a four-week, strengths-based leadership program.
  Two four-week leadership programs (15 youth per program) will be led by coaches from the research team's current TYOH 2.0 study with youth advisors participating as paid leadership interns.
  Interventions: Behavioral: Co-Designed Strengths-Based Leadership Program

INTERVENTIONS:
Behavioral: Co-Designed Strengths-Based Leadership Program — Please see arm description.

SUMMARY:
The idea for this study came from the research team's current study called Transitioning Youth Out of Homelessness (TYOH) 2.0, which provides coaching and a leadership guide to youth transitioning out of homelessness. Based on feedback from youth and coaches involved in that study, the research team plans to make small changes to the leadership guide and see if it works better as an in-person, four-week leadership program.

All participants in this study will be invited to attend an in-person, four-week leadership program. There will be two programs running at the same time: one in St. Catharines and one in Toronto. The goal is to have 15 participants in each program.

The main purpose of the study is to learn what participants think of the program. The second purpose is to see if there are changes in identity capital (feeling a sense of purpose and confidence in achieving goals) and knowledge about things that are covered in the program, when the research team compares participants' answers at the beginning and at the end of the program.

DETAILED DESCRIPTION:
This project builds on the research team's current community-based randomized clinical trial (Transitioning Youth Out of Homelessness 2.0) utilizing coaching and a co-designed leadership guide to target identity capital (purpose, control, self-efficacy, and self-esteem) for youth transitioning out of homelessness (all participants are also receiving rent subsidies). Based on preliminary feedback from study youth and coaches involved in the intervention arm, the research team will modify the leadership guide and pilot it in the form of an in-person, four-week leadership program (vs. independent learning in the current study).

The overarching objective of this mixed methods pilot project is to co-develop and test a strengths-based leadership program targeting identity capital for youth (16-24 years of age) transitioning out of homelessness. Specifically, the objectives are to:

1. Modify the leadership guide being used in the research team's current study so it can be delivered as an in-person leadership program.
2. Co-develop and pilot a four-week, strengths-based leadership program for young people transitioning out of homelessness.
3. Determine the feasibility and acceptability of the leadership guide when delivered as a four-week, in-person program (as opposed to independent learning in the current study).
4. Examine whether self-reported measures of identity capital and knowledge of program material show improvement immediately post-program compared to baseline.
5. Explore whether there are differences in outcomes by sub-groups (e.g., gender, age, identification as 2SLGBTQ+, child welfare involvement) and/or program participation levels.

If this modified delivery of the leadership guide shows promise, the research team plans to incorporate it into a national scale-up alongside rent subsidies and coaching.

ELIGIBILITY:
Eligible young people aged 16-24 years who have transitioned out of homelessness (e.g., no longer living in a shelter or couch surfing), defined as 3 consecutive months within the past 12 months, will be identified by community partners (note: for the purpose of this study, youth living in foster care will be considered homeless).

This age mandate was chosen because this is the age group served by the community partners. The research team has chosen to target the first year of exiting homelessness because collective experience has shown that this can be a particularly precarious time for youth in terms of mental health challenges and risk of (re)experiencing homelessness (even if youth have attempted exits in the past).

Inclusion Criteria:

* Be able to provide free and informed consent.
* Be able to understand English (leadership program and data collection will be conducted in English).
* Have experienced homelessness (e.g., unstable housing arrangements including shelter stays, foster care, and couch surfing) for 3 consecutive months in the past 12 months.
* Be able to consistently attend the four-week leadership program.

Exclusion Criteria:

* Enrolled in a program or study with similar features to the TYOH 2.5 leadership program.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Côté, J. (2016). The identity capital model: A handbook of theory, methods, and findings.
- See also: Describes the Multi-Measure Agentic Personality Scale (MAPS20), which is being utilized in the current study. — https://sociology.uwo.ca/research/research-areas/power-and-justice/Cote_ICM_Handbook_2016.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Leadership Program: Participants in this group participated in an in-person, four-week, strengths-based leadership program. The program was facilitated by professional coaches with youth advisors participating as paid leadership interns. The program consisted of eight 3-hour sessions and the curriculum aimed to improve identity capital (self-esteem, sense of purpose and control, self-efficacy).
Period: Overall Study
Arm/Group | Leadership Program
Started | 25
Completed | 18
Not Completed | 7
Not completed — Removed by study team | 2
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Leadership Program
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants] — Age categories reported at baseline: 16-18, 19-21, 22-24.
  Participants
    Age: 16-18 years | 6
    Age: 19-21 years | 10
    Age: 22-24 years | 9
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Boy/Man | 7
  Gender: Girl/Woman | 16
  Gender: Non-binary | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 7
  Race/Ethnicity: Black | 5
  Race/Ethnicity: Mixed | 8
  Race/Ethnicity: Other | 5
Sexual Orientation [Count of Participants; unit: Participants]
  Queer/gay/lesbian/bisexual/pansexual/questioning | 9
  Straight/heterosexual | 15
  Did not specify | 1
Immigration Status [Count of Participants; unit: Participants]
  Canadian Citizen | 19
  Permanent Resident | 5
  Refugee | 1
Child Welfare Involvement [Count of Participants; unit: Participants] — Participants were asked (self-report): "Has the Children's Aid Society (CAS) ever been involved with you or your family? (e.g., closely monitoring your well-being or moving you to foster care)"
  Participants
    Yes | 16
    No | 9
Age First Homeless [Count of Participants; unit: Participants]
  Before the age of 10 | 2
  10-12 years of age | 0
  13-15 years of age | 7
  16-18 years of age | 10
  19-21 years of age | 6
  22-25 years of age | 0
Attempts to Live on Own After Being Homeless [Count of Participants; unit: Participants]
  1-2 | 12
  3-4 | 11
  5 or more | 2
Highest Education Level [Count of Participants; unit: Participants]
  Less than grade 9 | 1
  Some high school | 11
  Completed high school | 7
  Some post-secondary (e.g., college, university, or vocational training after high school) | 5
  Completed post-secondary | 1
Regular Contact with Adult Relative [Count of Participants; unit: Participants] — Participants were asked (self-report): "Are you in regular contact with an adult relative? (e.g., parent, grandparent, or aunt)" Participants who chose not to answer this question are reported as "Did not specify."
  Participants
    Yes | 13
    No | 12
Adult that Provides Guidance and Encouragement [Count of Participants; unit: Participants] — Participants were asked (self-report): "Do you have an adult in your life who you are not related to that you can count on for guidance and encouragement?"
  Participants
    Yes | 17
    No | 8
Receiving Social Assistance [Count of Participants; unit: Participants] — Participants were asked (self-report): "Are you receiving OW, ODSP, or money from the Children's Aid Society (CAS)?" OW = Ontario Works; ODSP = Ontario Disability Support Program
  Participants
    Yes | 24
    No | 1
Access Food Assistance Programs [Count of Participants; unit: Participants]
  Yes | 13
  No | 12
Attending School (Secondary or Post-Secondary) [Count of Participants; unit: Participants]
  Yes | 11
  No | 13
  Did not specify | 1
Employed in Past Month [Count of Participants; unit: Participants]
  Yes | 6
  No | 18
  Did not specify | 1
Hours Worked Per Week in Past Month [Count of Participants; unit: Participants] — Population: This question was only asked of the participants who were employed in the past month (n = 6).
  Participants
    number analyzed (Participants) | 6
    1-20 | 3
    21-40 | 3
    Over 40 | 0
Job is Meaningful [Count of Participants; unit: Participants] — Participants were asked (self-report): "Is your job meaningful to you? (e.g., you enjoy it and/or it will help you achieve your life goals)" Population: This question was only asked of the participants who were employed in the past month (n = 6).
  Participants
    number analyzed (Participants) | 6
    Yes | 4
    No | 2
Participating in Training/Trades Program [Count of Participants; unit: Participants]
  Yes | 3
  No | 20
  Did not specify | 2

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility and Acceptability (Assessed by Recruitment/Enrolment/Completion Metrics)
Description: Quantitative measures consisting of recruitment/enrolment/completion metrics will be utilized.
  The recruitment rate will be estimated as the proportion of contacted individuals who express interest in participating in the study (T0).
  The enrolment rate will be calculated as the proportion of recruited individuals who are eligible and consent to participate in the study (T0).
  Participants were considered to have completed the study if they attended the final program session and completed final data collection (T2).
Time Frame: Assessed at T0 (pre-intervention), T1 (first day of intervention) and T2 (last day of intervention).
Population: Analysis population includes all participants screened for study eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Leadership Program
Number analyzed (Participants) | 35
Participants
  Screened | 35
  Enrolled | 25
  Completed Study | 18

2. Primary Outcome: Intervention Feasibility and Acceptability (Assessed by Program Attendance)
Description: Program attendance was calculated as the percentage of total possible leadership program sessions attended (maximum 8 sessions).
Time Frame: Assessed at T2 (last day of intervention).
Measure: Mean (Standard Deviation); unit: Percent of sessions attended
Arm/Group | Leadership Program
Number analyzed (Participants) | 25
Percent of sessions attended | 75.5 (20.9)

3. Primary Outcome: Intervention Feasibility and Acceptability (Assessed by Program Feedback Questionnaire)
Description: This 4-item anonymous questionnaire was developed for this study to collect information about participants' view of the leadership program, the impact of the program on them, and their view of the individuals running the program.
Time Frame: Assessed at T2 (last day of intervention).
Population: Analysis population includes participants who completed the study (i.e., attended the final program session and completed T2 data collection).
Measure: Count of Participants; unit: Participants
Arm/Group | Leadership Program
Number analyzed (Participants) | 18
Participants
  I would recommend this program to my friends or other youth I know with similar experiences.: Strongly disagree | 0
  I would recommend this program to my friends or other youth I know with similar experiences.: Disagree | 0
  I would recommend this program to my friends or other youth I know with similar experiences.: Slightly disagree | 0
  I would recommend this program to my friends or other youth I know with similar experiences.: Slightly agree | 1
  I would recommend this program to my friends or other youth I know with similar experiences.: Agree | 8
  I would recommend this program to my friends or other youth I know with similar experiences.: Strongly agree | 9
  The coaches and staff were knowledgeable about the program material.: Strongly disagree | 0
  The coaches and staff were knowledgeable about the program material.: Disagree | 0
  The coaches and staff were knowledgeable about the program material.: Slightly disagree | 0
  The coaches and staff were knowledgeable about the program material.: Slightly agree | 0
  The coaches and staff were knowledgeable about the program material.: Agree | 8
  The coaches and staff were knowledgeable about the program material.: Strongly agree | 10
  The coaches and staff were effective facilitators.: Strongly disagree | 0
  The coaches and staff were effective facilitators.: Disagree | 0
  The coaches and staff were effective facilitators.: Slightly disagree | 1
  The coaches and staff were effective facilitators.: Slightly agree | 0
  The coaches and staff were effective facilitators.: Agree | 7
  The coaches and staff were effective facilitators.: Strongly agree | 10
  Participating in this program has made a difference in my day-to-day life.: Strongly disagree | 0
  Participating in this program has made a difference in my day-to-day life.: Disagree | 1
  Participating in this program has made a difference in my day-to-day life.: Slightly disagree | 0
  Participating in this program has made a difference in my day-to-day life.: Slightly agree | 2
  Participating in this program has made a difference in my day-to-day life.: Agree | 5
  Participating in this program has made a difference in my day-to-day life.: Strongly agree | 10

4. Primary Outcome: Intervention Feasibility and Acceptability (Informed by Focus Groups)
Description: Focus group discussions (at T2) with program participants primarily centered around intervention acceptability but also explored the impact of the intervention on identity capital (e.g., sense of purpose and control) and socioeconomic inclusion (e.g., connection to broader social networks). Qualitative data analysis was conducted using reflexive thematic analysis with a critical social theoretical lens. During analysis, focus group transcripts were coded and codes were organized in a code book, clustered into categories, and eventually synthesized into key themes and sub-themes.
Time Frame: Assessed at T2 (last day of intervention).
Population: as for outcome 3
Measure: Number; unit: Themes
Arm/Group | Leadership Program
Number analyzed (Participants) | 18
Themes
  Key Themes | 3
  Sub-themes | 7

5. Secondary Outcome: Pre-post Intervention Change in Identity Capital (Assessed by Multi-Measure Agentic Personality Scale)
Description: The Multi-Measure Agentic Personality Scale (MAPS20) is a 20-item validated self-report measure that explores domains related to identity capital. The MAPS20 contains the following sub-scales: Self-Esteem; Purpose in Life; Internal Locus of Control; Self-Efficacy/Ego Strength. Each subscale has a score range of 5-30, with higher scores indicating greater identity capital.
Time Frame: Assessed at T1 (first day of intervention) and T2 (last day of intervention).
Population: T2 analysis population includes participants who completed the study (i.e., attended the final program session and completed T2 data collection).
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Leadership Program
Number analyzed (Participants) | 25
Score on a Scale
  Self-Esteem (T1) | 20.3 (4.0)
  Purpose in Life (T1) | 18.8 (4.8)
  Locus of Control (T1) | 20.8 (2.9)
  Self-Efficacy (T1) | 20.6 (4.0)
  Self-Esteem (T2): number analyzed (Participants) | 18
  Self-Esteem (T2) | 21.9 (4.4)
  Purpose in Life (T2): number analyzed (Participants) | 18
  Purpose in Life (T2) | 20.2 (5.4)
  Locus of Control (T2): number analyzed (Participants) | 18
  Locus of Control (T2) | 20.6 (3.8)
  Self-Efficacy (T2): number analyzed (Participants) | 18
  Self-Efficacy (T2) | 19.0 (4.2)
Statistical Analysis 1: Comparison: Leadership Program; Paired t-tests were conducted to compare T1 and T2 Self-Esteem (MAPS20 subscale) scores. This analysis included participants who completed both T1 and T2 data collection (n = 18); Test type: Other; p = 0.0011, t-test, 2 sided — Threshold for statistical significance: P <= 0.05. As this was an exploratory analysis only, p-values were not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Leadership Program; Paired t-tests were conducted to compare T1 and T2 Purpose in Life (MAPS20 subscale) scores. This analysis included participants who completed both T1 and T2 data collection (n = 18); Test type: Other; p = 0.0719, t-test, 2 sided — Threshold for statistical significance: P <= .05. As this was an exploratory analysis only, p-values were not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Leadership Program; Paired t-tests were conducted to compare T1 and T2 Locus of Control (MAPS20 subscale) scores. This analysis included participants who completed both T1 and T2 data collection (n = 18); Test type: Other; p = 0.7991, t-test, 2 sided — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: Leadership Program; Paired t-tests were conducted to compare T1 and T2 Self-Efficacy (MAPS20 subscale) scores. This analysis included participants who completed both T1 and T2 data collection (n = 18); Test type: Other; p = 0.2208, t-test, 2 sided — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: Leadership Program; We conducted an exploratory, descriptive analysis investigating the relationship between leadership program attendance and identity capital at T2, accounting for T1 scores (MAPS20 subscale: Self-Esteem). This analysis included participants who completed both T1 and T2 data collection (n = 18). We calculated the Spearman correlation coefficient only. Power calculation does not apply for this analysis; Test type: Other; Spearman partial correlation coefficient = 0.37
Statistical Analysis 6: Comparison: Leadership Program; We conducted an exploratory, descriptive analysis investigating the relationship between leadership program attendance and identity capital at T2, accounting for T1 scores (MAPS20 subscale: Purpose in Life). This analysis included participants who completed both T1 and T2 data collection (n = 18). We calculated the Spearman correlation coefficient only. Power calculation does not apply for this analysis; Test type: Other; Spearman partial correlation coefficient = -0.29
Statistical Analysis 7: Comparison: Leadership Program; We conducted an exploratory, descriptive analysis investigating the relationship between leadership program attendance and identity capital at T2, accounting for T1 scores (MAPS20 subscale: Locus of Control). This analysis included participants who completed both T1 and T2 data collection (n = 18). We calculated the Spearman correlation coefficient only. Power calculation does not apply for this analysis; Test type: Other; Spearman partial correlation coefficient = -0.58
Statistical Analysis 8: Comparison: Leadership Program; We conducted an exploratory, descriptive analysis investigating the relationship between leadership program attendance and identity capital at T2, accounting for T1 scores (MAPS20 subscale: Self-Efficacy). This analysis included participants who completed both T1 and T2 data collection (n = 18). We calculated the Spearman correlation coefficient only. Power calculation does not apply for this analysis; Test type: Other; Spearman partial correlation coefficient = -0.14

6. Secondary Outcome: Pre-post Intervention Change in Knowledge of Program Material
Description: The composite knowledge assessment scale is 16-item self-report measure that was developed for this study and explores concepts from the program curriculum, such as: mindfulness; core values; purpose; goal setting; growth mindset; identity; and courage. Reported values represent the percentage of participants who answered the question correctly (i.e., agreeing with a correct statement or disagreeing with an incorrect statement).
Time Frame: Assessed at T1 (first day of intervention) and T2 (last day of intervention).
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Leadership Program
Number analyzed (Participants) | 25
Percentage of participants
  I am confident about my ability to be in the driver's seat in my "car of life." (T1) | 76.0
  I can name at least one strategy that I consistently use to help me accomplish my daily tasks. (T1) | 88.0
  It is more important to focus on what you want to achieve than who you wish to become. (T1) | 40.0
  I have a good understanding of how my brain becomes anxious. (T1) | 87.5
  I am confident in my purpose and why it is important in my life. (T1) | 80.0
  People who believe they are worthy of love/belonging have an easier time showing vulnerability. (T1) | 100.0
  I am not very confident about knowing how to get my "wise mind" in control. (T1) | 52.0
  I have a good understanding of how to create an environment that helps me achieve my goals. (T1) | 84.0
  I have a hard time naming things around me that have contributed to my habits. (T1) | 56.0
  I am confident that I have the knowledge/skills to "speak back" to feelings of shame. (T1) | 76.0
  I can easily name my core values. (T1) | 84.0
  When creating a new habit (e.g., exercising) it is important to stop while it still feels good. (T1) | 41.7
  Your intelligence is something very basic about you that you can't change very much. (T1) | 72.0
  It is more important to strive for excellence than perfection. (T1) | 84.0
  You need to connect with others before you can connect with yourself. (T1) | 62.5
  Interdependence is an important part of self-leadership. (T1) | 87.5
  I am confident about my ability to be in the driver's seat in my "car of life." (T2): number analyzed (Participants) | 18
  I am confident about my ability to be in the driver's seat in my "car of life." (T2) | 83.3
  I can name at least one strategy that I consistently use to help me accomplish my daily tasks. (T2): number analyzed (Participants) | 18
  I can name at least one strategy that I consistently use to help me accomplish my daily tasks. (T2) | 94.4
  It is more important to focus on what you want to achieve than who you wish to become. (T2): number analyzed (Participants) | 18
  It is more important to focus on what you want to achieve than who you wish to become. (T2) | 29.4
  I have a good understanding of how my brain becomes anxious. (T2): number analyzed (Participants) | 18
  I have a good understanding of how my brain becomes anxious. (T2) | 100.0
  I am confident in my purpose and why it is important in my life. (T2): number analyzed (Participants) | 18
  I am confident in my purpose and why it is important in my life. (T2) | 94.4
  People who believe they are worthy of love/belonging have an easier time showing vulnerability. (T2): number analyzed (Participants) | 18
  People who believe they are worthy of love/belonging have an easier time showing vulnerability. (T2) | 83.3
  I am not very confident about knowing how to get my "wise mind" in control. (T2): number analyzed (Participants) | 18
  I am not very confident about knowing how to get my "wise mind" in control. (T2) | 55.6
  I have a good understanding of how to create an environment that helps me achieve my goals. (T2): number analyzed (Participants) | 18
  I have a good understanding of how to create an environment that helps me achieve my goals. (T2) | 88.9
  I have a hard time naming things around me that have contributed to my habits. (T2): number analyzed (Participants) | 18
  I have a hard time naming things around me that have contributed to my habits. (T2) | 83.3
  I am confident that I have the knowledge/skills to "speak back" to feelings of shame. (T2): number analyzed (Participants) | 18
  I am confident that I have the knowledge/skills to "speak back" to feelings of shame. (T2) | 82.4
  I can easily name my core values. (T2): number analyzed (Participants) | 18
  I can easily name my core values. (T2) | 100.0
  When creating a new habit (e.g., exercising) it is important to stop while it still feels good. (T2): number analyzed (Participants) | 18
  When creating a new habit (e.g., exercising) it is important to stop while it still feels good. (T2) | 72.2
  Your intelligence is something very basic about you that you can't change very much. (T2): number analyzed (Participants) | 18
  Your intelligence is something very basic about you that you can't change very much. (T2) | 32.2
  It is more important to strive for excellence than perfection. (T2): number analyzed (Participants) | 18
  It is more important to strive for excellence than perfection. (T2) | 94.4
  You need to connect with others before you can connect with yourself. (T2): number analyzed (Participants) | 18
  You need to connect with others before you can connect with yourself. (T2) | 77.8
  Interdependence is an important part of self-leadership. (T2): number analyzed (Participants) | 18
  Interdependence is an important part of self-leadership. (T2) | 88.9

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Leadership Program
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
This is a feasibility and acceptability study and thus not adequately powered to detect a significant difference in quantitative self-report measures; results must be interpreted with caution. All young people will be connected to urban-based social service agencies in the province of Ontario; other youth populations may differ. Quantitative instruments are based on self-reports and thus subject to social desirability bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT06425458/Prot_SAP_000.pdf